CLINICAL TRIAL: NCT05451186
Title: The Effect of Eye Patch and Headset on Sleep Quality, Anxiety, Fear and Vital Signs in Intensive Care Patients: A Randomized Controlled Study
Brief Title: The Eye Patch and Headset on Sleep Quality, Anxiety, Fear and Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8991
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Intensive Care Unit; Headphones; Sleep bands; Sleep

STUDY DESIGN:
Intervention Model Description: This research is a single-blind study with a pretest-posttest randomized control group.
Who Masked: Participant
Masking Description: Experimental group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye patch and headphones (Experimental): Eye patch and headphones
  Interventions: Other: Eye patch and headphones
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Eye patch and headphones — Patients in the experimental group will be asked to use an eye mask and earplugs from 22:30 to 6:30 in the morning on the 1st, 2nd and 3rd nights.
  Arms: Eye patch and headphones

SUMMARY:
This study was planned to investigate the effects of eye patch and headphones on sleep quality, anxiety, fear and vital signs in coronary intensive care unit patients.

DETAILED DESCRIPTION:
In intensive care units, it can be much easier to change the environment perception of patients with simple tools such as headphones and sleep bands, rather than changing the environment of the patients. The use of sleep bands and headphones, which are non-pharmacological methods, can reduce sleep deprivation by changing the environmental perception of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* New York Heart Association (NYHA) functional class II and III,
* Not having received any general anaesthesia for the previous 24 hours,
* Not having received any sedative medications or opioids for the past 24 hours,
* Not having a verbal communication disability (hearing and speaking),
* Absence of pain,
* Not having a previously diagnosed sleep disorder,
* Not having psychiatric problems,
* Not having a cognitive problem,
* Being healthy enough to put on and take off earplugs independently, in addition to wearing an eye mask and removing it when necessary, and continuing to be hospitalized for at least three days.

Exclusion Criteria:

* Diagnosed with delirium (Intensive care delirium screening checklist >=5),
* Unconscious (Glasgow coma scale<13),
* Presence of additional chronic diseases,
* Having consumed coffee, alcohol and hypnotic drugs at least 12 hours before the study,
* Patients whose condition suddenly worsened,
* Those who cannot use earplugs and eye masks effectively at night,
* Those who voluntarily withdrew from the study and were transferred from the intensive care unit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (Fear) | the first day after receiving randomisation
  Patients are asked to show the severity of their fear on a 10 cm long vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale (Anxiety) | the first day after receiving randomisation
  Patients are asked to show the severity of their anxiety on a 10 cm long vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Vital Signs Follow-up Form | the first day after receiving randomisation
  This form was created by the researcher in order to record the systolic-diastolic blood pressure, and heart rate (pulse), values of the patient who was applied an eye patch or earphone at night.
The Richards-Campbell Sleep Questionnaire | the first day after receiving randomisation
  This brief five-item questionnaire was used to evaluate perceived sleep depth, sleep latency (time to fall asleep), number of awakenings, efficiency (percentage of time awake), and sleep quality. It also includes a sixth item evaluating perceived night-time noise. Each item is evaluated on a scale of 0-100 with a visual analogue scale technique. A score of 0-25 indicates very poor quality sleep, whereas a score of 76-100 indicates very good sleep quality.

SECONDARY OUTCOMES:
Visual Analog Scale (Fear) | 4. days
  Patients are asked to show the severity of their fear on a 10 cm long vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale (Anxiety) | 4. days
  Patients are asked to show the severity of their anxiety on a 10 cm long vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Vital Signs Follow-up Form | 4. days
  This form was created by the researcher in order to record the systolic-diastolic blood pressure, and heart rate (pulse), values of the patient who was applied an eye patch or earphone at night.
The Richards-Campbell Sleep Questionnaire | 4. days
  This brief five-item questionnaire was used to evaluate perceived sleep depth, sleep latency (time to fall asleep), number of awakenings, efficiency (percentage of time awake), and sleep quality. It also includes a sixth item evaluating perceived night-time noise. Each item is evaluated on a scale of 0-100 with a visual analogue scale technique. A score of 0-25 indicates very poor quality sleep, whereas a score of 76-100 indicates very good sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, Study Director — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kasapoglu ES, Enc N. Role of multicomponent non-pharmacological nursing interventions on delirium prevention: A randomized controlled study. Geriatr Nurs. 2022 Mar-Apr;44:207-214. doi: 10.1016/j.gerinurse.2022.02.015. Epub 2022 Feb 26. PMID 35227973